CLINICAL TRIAL: NCT04510610
Title: An Open-label, Multicenter, phase2/3 Study of Camrelizumab Plus Decitabine in Anti-PD-1 Treatment-naive Patients With Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Camrelizumab Plus Decitabine in Anti-PD-1 Treatment-naive Patients With Relapsed/Refractory Classical Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-056
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — camrelizumab; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab plus decitabine (Experimental): Decitabine 10 mg/day, days 1-5; Camrelizumab 200 mg, day 8, every 3 weeks.
  Interventions: Drug: Camrelizumab and Decitabine

INTERVENTIONS:
Drug: Camrelizumab and Decitabine — Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1 (DNMT1), which can increase tumor antigens and HLA expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function. Camrelizumab is a humanized anti-PD-1 monoclonal antibody.

SUMMARY:
This is an open-label, Phase 2/3，multicenter and single-arm clinical trial of Camrelizumab plus decitabine for Anti-PD-1 treatment-naive patients with relapsed or refractory Hodgkin Lymphoma. The primary objective of this study is to evaluate the long-term response duration with Camrelizumab plus decitabine in relapsed or refractory Hodgkin Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1 Subjects must have histological confirmation of relapsed or refractory Hodgkin lymphoma (HL).
* 2 12 to 75 years of age.
* 3 ECOG performance of less than 2.
* 4 Life expectancy of at least 3 months.
* 5 Subjects with lymphoma must have at least one measureable lesion >1 cm as defined by lymphoma response criteria.
* 6 Subjects must have received at least two lines of prior regimens without Anti-PD-1 antibody treatment history, and must be off therapy for at least 4 weeks prior to Day 1. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months.
* 7 Subjects must have adequate marrow, live, renal and heart functions.

Exclusion Criteria:

* 1 Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
* 2 Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
* 3 Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in 1 month .
* 4 Prior organ allograft.
* 5 Women who are pregnant or breastfeeding.
* 6 Women with a positive pregnancy test on enrollment or prior to nvestigational product administration.
* 7 Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
duration of response | 5 years
  Time measured from the day of first documented PR or CR to the date of first documented progression, or death from any cause.
Progression free survival | 5 years
  Time measured from the day of treatment to the date of first documented progression, or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Hematology Department of Chinese PLA General Hospital, Beijing, China